CLINICAL TRIAL: NCT03327428
Title: Register Sichelzellkrankheit Der GPOH
Brief Title: Sickle-cell Disease Registry of the GPOH
Acronym: SichReg
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: GPOH Consortium Sickle Cell Disease (Other); Johann Wolfgang Goethe University Hospital (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Ulm (Other); Charite University, Berlin, Germany (Other); German Cancer Research Center (Other); Deutsche Kinderkrebsstiftung (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Joachim Kunz, Senior physician, University Hospital Heidelberg
Other Study IDs: Register Sichelzellkrankheit
Record Dates: First submitted 2017-08-16; First posted 2017-10-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease
Keywords: Anemia, Sickle Cell; Sickle Cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Sickle Cell Disease: Patients with any sickling condition, including among others Sickle Cell Anemia, HbSC Disease, HbS-betaThal, excluding Sickle Cell Trait.

SUMMARY:
Sickle cell disease is one of the most common hereditary diseases. Most severe complications can be avoided if the disease is detected early and treated appropriately.

The sickle cell disease registry of the Society for Paediatric Oncology/Haematology aims at describing the epidemiology of sickle cell disease in German-speaking central Europe. Patients with sickle cell disease will be characterized clinically and genetically and treatment will be documented with the aim to find predictors of the course of disease.

In addition, the registry results should provide a solid evidence base to incorporate sickle cell disease into routine newborn screening and to update the national guidelines for the management of patients suffering from sickle cell disease in Germany.

A consortium of five university hospitals (Berlin, Frankfurt, Hamburg, Heidelberg, Ulm) has been mandated by the Society for Paediatric Oncology/Haematology to implement this registry.

The number of participating centers is constantly increasing and new centers that take care of either pediatric or adult patients with sickle cell disease are encouraged to support the registry.

For further information please refer to: http://www.sichelzellkrankheit.info/

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* current residency in either Germany, Austria or Switzerland
* sickle cell disease confirmed by hemoglobin analysis or molecular genetic analysis

  * Homozygous sickle cell disease (HbSS)
  * HbSC disease
  * Sickle cell disease HbS / bThal
  * Other, rare sickle cell syndromes such as HbS/OArab, HbS/HPFH, HbS/E, HbS/D Punjab, HbS/C Harlem, HbC/S Antilles, HbS/Quebec-CHORI, HbA/S Oman, HbA/Jamaica Plain

Exclusion Criteria:

- isolated heterozygous trait for HbS

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with sickle cell disease being treated at participating centers that signed the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in incidence of sickle-cell disease | Baseline and yearly, up to 10 years
  The incidence of sickle-cell disease will be reported every year in comparison to the preceding Report.

SECONDARY OUTCOMES:
Complications of sickle-cell disease | Baseline and yearly, up to 10 years
  In addition to the incidence of the disease itself also possible complications will be reported in comparison to the preceding report (in case of the first report, only the prevalence will be reported as baseline).
Treatment of sickle-cell disease | Baseline and yearly, up to 10 years
  In addition to the incidence of the disease itself also the treatment received will be reported in comparison to the preceding report (in case of the first report, only the prevalence will be reported as baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Kunz, Dr., Principal Investigator — Center for Child and Adolescent Medicine, University Medical Center Heidelberg; Holger Cario, Prof. Dr. — University Hospital Ulm; Regine Grosse, Dr.; Andrea Jarisch, Dr. — Johann Wolfgang Goethe University Hospital; Andreas Kulozik, Prof. Dr. — University Hospital Heidelberg; Stephan Lobitz, Dr. MSc — Gemeinschaftsklinikum Mittelrhein, Koblenz; Lena Oevermann — Charite University, Berlin, Germany
Locations (1):
- Center for Child and Adolescent Medicine, University Medical Center Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobitz S. Neugeborenenscreening auf Sichelzellkrankheiten in Deutschland. Kinder- und Jugendmedizin 2017;17(2):82-86 [German]
- [Background] Kunz JB, Cario H, Grosse R, Jarisch A, Lobitz S, Kulozik AE. The epidemiology of sickle cell disease in Germany following recent large-scale immigration. Pediatr Blood Cancer. 2017 Jul;64(7). doi: 10.1002/pbc.26550. Epub 2017 Apr 6. PMID 28383793
- [Background] Kunz JB, Awad S, Happich M, Muckenthaler L, Lindner M, Gramer G, Okun JG, Hoffmann GF, Bruckner T, Muckenthaler MU, Kulozik AE. Significant prevalence of sickle cell disease in Southwest Germany: results from a birth cohort study indicate the necessity for newborn screening. Ann Hematol. 2016 Feb;95(3):397-402. doi: 10.1007/s00277-015-2573-y. Epub 2015 Dec 12. PMID 26658910
- [Background] Grosse R, Lukacs Z, Cobos PN, Oyen F, Ehmen C, Muntau B, Timmann C, Noack B. The Prevalence of Sickle Cell Disease and Its Implication for Newborn Screening in Germany (Hamburg Metropolitan Area). Pediatr Blood Cancer. 2016 Jan;63(1):168-70. doi: 10.1002/pbc.25706. Epub 2015 Aug 14. PMID 26275168
- [Background] Frommel C, Brose A, Klein J, Blankenstein O, Lobitz S. Newborn screening for sickle cell disease: technical and legal aspects of a German pilot study with 38,220 participants. Biomed Res Int. 2014;2014:695828. doi: 10.1155/2014/695828. Epub 2014 Jul 23. PMID 25147811
- [Background] Lobitz S, Frommel C, Brose A, Klein J, Blankenstein O. Incidence of sickle cell disease in an unselected cohort of neonates born in Berlin, Germany. Eur J Hum Genet. 2014 Aug;22(8):1051-3. doi: 10.1038/ejhg.2013.286. Epub 2014 Jan 8. PMID 24398797
- [Result] Kunz JB, Lobitz S, Grosse R, Oevermann L, Hakimeh D, Jarisch A, Cario H, Beier R, Schenk D, Schneider D, Gross-Wieltsch U, Prokop A, Heine S, Khurana C, Erlacher M, Durken M, Linke C, Fruhwald M, Corbacioglu S, Claviez A, Metzler M, Ebinger M, Full H, Wiesel T, Eberl W, Reinhard H, Tagliaferri L, Allard P, Karapanagiotou-Schenkel I, Rother LM, Beck D, Le Cornet L, Kulozik AE; German Sickle Cell Disease Registry. Sickle cell disease in Germany: Results from a national registry. Pediatr Blood Cancer. 2020 Apr;67(4):e28130. doi: 10.1002/pbc.28130. Epub 2019 Dec 22. PMID 31867835
- [Result] Kunz JB, Schlotmann A, Daubenbuchel A, Lobitz S, Jarisch A, Grosse R, Cario H, Oevermann L, Hakimeh D, Tagliaferri L, Kulozik AE. Benefits of a Disease Management Program for Sickle Cell Disease in Germany 2011-2019: The Increased Use of Hydroxyurea Correlates with a Reduced Frequency of Acute Chest Syndrome. J Clin Med. 2021 Sep 30;10(19):4543. doi: 10.3390/jcm10194543. PMID 34640578
- [Result] Allard P, Alhaj N, Lobitz S, Cario H, Jarisch A, Grosse R, Oevermann L, Hakimeh D, Tagliaferri L, Kohne E, Kopp-Schneider A, Kulozik AE, Kunz JB. Genetic modifiers of fetal hemoglobin affect the course of sickle cell disease in patients treated with hydroxyurea. Haematologica. 2022 Jul 1;107(7):1577-1588. doi: 10.3324/haematol.2021.278952. PMID 34706496
- See also: Official website of the Registry [German] — http://www.sichelzellkrankheit.info/
- See also: Sickle Cell Disease Guidelines, German language — https://www.awmf.org/leitlinien/detail/ll/025-016.html